CLINICAL TRIAL: NCT03348254
Title: Single Shot Versus Multiple Shot Antibiotic Prophylaxis in Primary Joint Arthroplasty of the Hip and Knee, Comparison of Different Prophylaxis Regimes on the Risk of Revision for Infection
Brief Title: Antibiotic Prophylaxis in Primary Joint Arthroplasty of the Hip and Knee.
Status: Completed | Type: Observational
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Principal Investigator, Rudolf W Poolman, MD PhD, MD PhD, Orthopaedic surgeon, Onze Lieve Vrouwe Gasthuis
Other Study IDs: OLVG AB Profylaxe Veltman
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee; Antibiotic Prophylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Group one will consist of patients receiving a single shot antibiotic prophylaxis preoperatively before primary arthroplasty of hip or knee
  Interventions: Drug: Single shot antibiotic prophylaxis
- 2: Group two will consist of patients receiving multiple shot antibiotic prophylaxis perioperatively before and after primary arthroplasty of hip or knee
  Interventions: Drug: Multiple shot antibiotic prophylaxis

INTERVENTIONS:
Drug: Single shot antibiotic prophylaxis — single shot preoperative antibiotic prophylaxis
  Groups: 1
Drug: Multiple shot antibiotic prophylaxis — Multiple shot perioperative antibiotic prophylaxis
  Groups: 2

SUMMARY:
A retrospective study will be performed to compare the incidence of revision procedures performed for the treatment of postoperative periprosthetic joint infection (PJI) between patients treated with a single preoperative antibiotic prophylaxis and patients treated with multiple shot antibiotic prophylaxis following primary arthroplasty of hip or knee.

This study will be conducted in two phases. In phase 1 the investigators will evaluate which antibiotic prophylaxes (type of antibiotic and duration of prophylaxis) are regularly used in the Netherlands, by contacting all orthopaedic centres implanting total hip and total knee prostheses. In phase 2 the investigators will compare infection rate (defined as revision for infection as registered in the LROI database) between a single-shot and multiple shot antibiotic prophylaxis.

Knee and hip primary arthroplasties will be considered separately.

DETAILED DESCRIPTION:
In phase 1 of this study all Dutch hospitals and clinics performing hip and/or knee arthroplasty will be contacted to supply data concerning type and duration of antibiotic prophylaxis. The investigators will also ask whether debridement with implant retention for early infection is registered in the LROI. The investigators will ask permission to have access to unblended data on institutional level to be able to connect the type of antibiotic prophylaxis to outcome.

In phase 2 the investigators will include all adult patients whom have a primary hip or knee arthroplasty and are registered in the national joint implant registry (LROI) between 2011 and 2016.Those patients will be followed until they are revised (irrespectively of the indication), they died or the end-point of the study, i.e. end of 2016 (to allow at least one year follow-up for those operated late 2015).

Exclusion criteria are patients aged under 18. Patients with no primary procedure recorded in the LROI for the period of interest but records of revision surgeries will be excluded.

The investigators will compare the results found in the LROI database in two groups for both hip and knee arthroplasties. Group one will consist of patients receiving a single shot antibiotic prophylaxis, while group two will consist of patients receiving multiple shot antibiotic prophylaxis.

Analyses will be adjusted for known and available confounders such as age, gender, BMI, and ASA score.

In the LROI debridement without exchange of mobile parts for early infection, is only scarcely reported. The authors realise not all early infection treatments, such as debridement with or without exchange of mobile parts, are registered in the LROI database.

ELIGIBILITY:
Inclusion Criteria:

- All adult patients whom have a primary hip or knee arthroplasty and are registered in the national joint implant registry (LROI) between 2011 and 2014

Exclusion Criteria:

* Patients aged under 18.
* Patients with no primary procedure recorded in the LROI for the period of interest but records of revision surgeries will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients whom have a primary hip or knee arthroplasty and are registered in the national joint implant registry (LROI) between 2011 and 2014. Those patients will be followed until they are revised (irrespectively of the indication), they died or the end-point of the study, i.e. end of 2015 (to allow at least one year follow-up for those operated late 2014).
Sampling Method: Probability Sample
Enrollment: 242179 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Revision arthroplasty because of infection | one year
  Revision of the hip or knee prosthesis because of infection within one year after primary surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf W Poolman, MD PhD, Principal Investigator — OLVG
Locations (1):
- OLVG, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veltman ES, Lenguerrand E, Moojen DJF, Whitehouse MR, Nelissen RGHH, Blom AW, Poolman RW. Similar risk of complete revision for infection with single-dose versus multiple-dose antibiotic prophylaxis in primary arthroplasty of the hip and knee: results of an observational cohort study in the Dutch Arthroplasty Register in 242,179 patients. Acta Orthop. 2020 Dec;91(6):794-800. doi: 10.1080/17453674.2020.1794096. Epub 2020 Jul 23. PMID 32698642